CLINICAL TRIAL: NCT04768582
Title: Platelet Reactivity After an Eastern Asian Loading Dose of Prasugrel in Taiwanese Patients With Acute Myocardial Infarction: PREP-TAMI Study
Brief Title: Platelet Reactivity After an Eastern Asian Loading Dose of Prasugrel in Taiwanese ACS Patients
Acronym: PREP-TAMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Feng Yuan Hospital, Ministry of Health and Welfare (Other Government)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Chen-Rong, Tsao M.D., Chief of Cardiology, Feng Yuan Hospital, Ministry of Health and Welfare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FYHIRB109001
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Acute Coronary Syndrome; Hemorrhage; Treatment Side Effects
Keywords: Acute Coronary Syndrome; Prasugrel; VerifyNow-P2Y12 assay
MeSH Terms: conditions — Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efient group (Experimental): ACS patients who received oral Prasugrel after coronary angiography been done
  Interventions: Diagnostic Test: P2Y12-reaction-units (PRU) by VerifyNow-P2Y12 assay

INTERVENTIONS:
Diagnostic Test: P2Y12-reaction-units (PRU) by VerifyNow-P2Y12 assay — The efficacy endpoint was platelet reactivity, of which was serially assessed using the VerifyNow-P2Y12 assay and the results were expressed as P2Y12-reaction-units (PRU).

SUMMARY:
Prasugrel has a faster onset of action and greater platelet inhibition with less inter-individual response variability than clopidogrel. Japan and Taiwan are the only two nations where adjusted/Asian dose of prasugrel (loading dose (LD)/maintenance (MD): 20/3.75 mg) was approved for clinical use. However, there is no data regarding the effectiveness of adjusted dose of prasugrel on platelet reactivity in Taiwanese patients with acute coronary syndrome (ACS). This study aim to evaluate the pharmacodynamic of the Asian dose prasugrel on the platelet reactivity after percutaneous coronary intervention (PCI) for patients with ACS.

DETAILED DESCRIPTION:
Rationale and Background Prasugrel provides more potent and rapid platelet inhibition compared to Clopidogrel.

Rapid and effective inhibition of the platelet P2Y12 receptor is of pivotal importance in patients with AMI who undergo PCI.

Prasugrel (60 mg loading and 10 mg/day maintenance dose) is a new generation P2Y12 inhibitor that achieves greater and faster platelet inhibition comparing with clopidogrel in patients undergoing PCI.

As revealed by 2 head-to-head studies, reducing Prasugrel dosages to 20/3.75 LD/MD (mg) was still efficacious but led to less bleeding events than the original 60/10 LD/MD (mg).

In TRITON-TIMI 38 trial, prasugrel was associated with not only significantly less ischemic events but also more non-CABG TIMI major bleeding, as compared to Clopidogrel.

In the PRASFIT-ACS study from Japan (20 mg loading and 3.75 mg/day maintenance dose), prasugrel was associated with a 23% reduction of MACE and the incidence of non-CABG major bleeding was similar to clopidogrel.

There is NO data regarding the effectiveness of Japanese loading dose of prasugrel on platelet reactivity in Taiwanese patients with AMI.

This study use PRU for efficacy and ISTH major bleeding for safety evaluations; the anticipated results are prompt and effective platelet inhibition as well as comparably low bleeding rate.

ELIGIBILITY:
Inclusion Criteria:

* Age>=20
* Mentally competent to provide an informed consent.
* A person being diagnosed with acute coronary syndrome and arranged for a percutaneous coronary intervention.

Exclusion Criteria:

* A history of hemorrhagic stroke at any time in the past.
* Active internal bleeding or has a history of a bleeding disorder (i.e. hemophilia).
* Severe liver disease; for example, cirrhosis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
platelet reactivity (PRU) after loading of prasugrel at 12 hours | 12 hours
  PRU 12 hours after a loading dose

SECONDARY OUTCOMES:
platelet reactivity (PRU) after loading of prasugrel at 1 hour | one hour
  PRU 1 hour after a loading dose
platelet reactivity (PRU) after loading of prasugrel at 3 hours | 3 hours
  PRU 3 hours after a loading dose
platelet reactivity (PRU) after loading of prasugrel at 48 hours | 48 hours
  PRU 48 hours after a loading dose
ISTH Major bleeding | day 7 after a loading dose of prasugrel
  the definition recommended by the International Society on Thrombosis and Haemostasis (ISTH) defines major bleeding as fatal bleeding; symptomatic bleeding in a critical area or organ such as intracranial, intraspinal, intraocular resulting in vision changes, retroperitoneal, intraarticular, pericardial

CONTACTS AND LOCATIONS:
Overall Officials: CHEN RONG TSAO, M.D., Principal Investigator — Feng Yuang Hospital
Locations (1):
- Feng Yuan Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No